CLINICAL TRIAL: NCT04989725
Title: Stereotactic Ablative Radiotherapy for Oligo-Progressive Disease REfractory to Systemic Therapy in Metastatic Cancer: A Phase II Randomized Trial
Brief Title: Stereotactic Ablative Radiotherapy for Oligo-Progressive Disease REfractory to Systemic Therapy in Metastatic Cancer
Acronym: SUPPRESS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Suppress
Record Dates: First submitted 2021-07-30; First posted 2021-08-04 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Head and Neck Cancer; Metastatic Cancer; Oligoprogressive
Keywords: head and neck cancer; metastatic cancer; oligoprogression
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Randomized screening phase II trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Switch to subsequent systemic therapy line, best supportive care or continue current systemic line
  Interventions: Other: Standard arm
- Experimental SABR arm (Experimental): Definitive SABR to oligoprogressive lesions + continue current systemic therapy
  Interventions: Radiation: Experimental arm

INTERVENTIONS:
Other: Standard arm — Patients on the standard arm will be treated as per standard of care in our institution. Treatment options could include switching to next systemic therapy line, best supportive care or continuing on current systemic therapy.
  Arms: Standard of care
Radiation: Experimental arm — SABR to all oligoprogressive lesions + continuation of current systemic therapy
  Arms: Experimental SABR arm

SUMMARY:
A registry-based randomized phase II trial. A total of 46 patients with metastatic head and neck cancer on systemic therapy with oligoprogression to 1-5 extracranial lesions will be randomized using a 1:1 ratio to standard of care (begin next-line systemic therapy, best supportive care, continue current systemic line, based on treating physician decision) vs. receive stereotactic ablative radiotherapy to all oligoprogressive lesions while continuing their current systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Biopsy proven HNSCC (oropharynx, oral cavity, nasopharynx, sinonasal, larynx or hypopharynx)
* Metastatic HNSCC, with pathological or radiological proof of metastasis
* Ability to provide written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Progressive disease while on systemic treatment (any line), defined as per RECIST criteria 1.1 on CT metrics as a greater than 20% increase in the sum measurement of lesions, non-target unequivocal progressive disease or a new lesion on CT.
* Oligoprogression to 1-5 extracranial lesions ≤ 5cm and involving ≤ 3 organs. Progression at the primary tumor site should be counted within the total of 5 lesions. For patients with lymph node metastases, each node is counted as one site of metastasis.
* All sites of disease can, in the opinion of the investigator, be safely treated and targetable with SABR (taking into account prior local therapy, organ function and underlying medical condition such as inflammatory bowel disease, pulmonary fibrosis, etc.)
* Patients with prior metastases that have been treated with ablative therapies (e.g. radiotherapy, surgery or radiofrequency ablation) before their current line of systemic therapy, are eligible.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Any medical condition that could, in the opinion of the investigator, preclude radiotherapy or prevent follow-up after radiotherapy.
* Presence of spinal cord compression
* Metastatic disease that invades the GI tract (including esophagus, stomach, small or large bowel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 5 years
  PFS defined from randomization to disease progression at any site or death

SECONDARY OUTCOMES:
Overall survival | 5 years
  OS defined as time from randomization to time of death from any cause.
Quality of life Measured using the FACT-G tool, head and neck cancer-related patient reported outcome- CTCAE (PRO-CTCAE) and Quality of life 5-level EQ-5D | 5 years
  Measured using the FACT-G tool, lung cancer-related patient reported outcome- CTCAE (PRO-CTCAE) and quality of life 5-level EQ-5D
Grade ≥ 3 toxicity Measured using the Common Terminology Criteria for Adverse Events (CTCAE v5.0) | 5 years
  Measured using the Common Terminology Criteria for Adverse Events
Local control | 5 years
  Defined as time from the end of SABR treatment to date of local failure and will be measured only in the experimental arm
Time to next systemic therapy | 5 years
  Defined as time from randomization to time of subsequent therapy line

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No